CLINICAL TRIAL: NCT06912893
Title: Efficacy of Radial and Focused Extracorporeal Shockwave Therapy in Patients Wirh Carpal Tunnel Syndrom. a Multicentric, Randomised Observer-blinded Trial
Brief Title: Clinical Efficiency Testing of Extracorporeal Radial and Focused Shock Wave Therapy in Patients With Mild to Moderate Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital St. Polten (Other)
Responsible Party: Principal Investigator, Dr. Constantin Dolle, Dr. med. univ., University Hospital St. Polten
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GS3-EK-1/222-2024
Record Dates: First submitted 2025-03-21; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- focused shockwave therapy (Active Comparator): this arm includes 30 patients with mild to moderate carpal tunnel syndrom who will receive therapy with focused shockwave therapy
  Interventions: Device: focused shock wave therapy
- radial shockwave therapy (Active Comparator): this arm includes 30 patients with mild to moderate carpal tunnel syndrom who will receive therapy with radial shockwave therapy
  Interventions: Device: radial shock wave therapy

INTERVENTIONS:
Device: radial shock wave therapy — treatment of the nervus medianus on the level of the carpal tunnel with radial shock wave therapy with 1500 impulses, 5 Hz and 1,5 bar
  Arms: radial shockwave therapy
Device: focused shock wave therapy — treatment of the nervus medianus on the level of the carpal tunnel with focused shock wave therapy with 1500 impulses, 5 Hz and 0,05 mJ/mm²
  Arms: focused shockwave therapy

SUMMARY:
The aim of the project is to test the efficacy of extracorporeal shock wave therapy (radial + focused) on clinical outcomes in patients with carpal tunnel syndrome (CTS). Shock wave therapy has already been shown to be potentially effective in the literature. However, no studies are known to date that test both shock wave types in one protocol, and the follow-up period in the previous studies was set at a maximum of 24 weeks.

Consequently, this study is planned as a multicenter, prospective, randomized, investigator-blinded study. 60 subjects will be assigned to the two shock wave types, and the follow-up period is scheduled for 32 weeks.

The study will be conducted at the Institute for Physical Medicine and Rehabilitation at the University Hospital Krems and St. Pölten. Recruitment will take place through the respective CTS outpatient clinics of the departments, as well as through private practice (orthopedists, general practitioners, neurologists, etc.). The inclusion and exclusion criteria are checked before the subject is included in the study, with nerve conduction velocity (NCV) being emphasized as a diagnostic method.

After the patient is included in the study or signs the consent form, the relevant demographic, medical, and personal data are collected (pseudonymized procedure). Study-related measurements are then performed (nerve sonography, Boston Carpal Tunnel Questionnaire, Visual Analog Scale). The baseline examinations and follow-up examinations are each performed by the same physician (blinded), while the subsequent shock wave therapy is performed by a second physician.

After the baseline examinations, the patient is randomly assigned to one of the two shock wave groups and receives five shock wave therapy sessions one week apart. The pulses and frequency of both treatments are identical (2000 and 5 Hz, respectively). The intensity is xx bar in the radial group and 0.05 mj/mm² in the focused group.

Detailed follow-up assessments, including all baseline measurements, will be conducted 16 and 32 weeks after the first shock wave therapy. At weeks 8 and 24, a questionnaire (Boston Carpal Tunnel Questionnaire; VAS) will also be sent to the patient.

Patients with bilateral clinical CTS will serve as the control group. In this case, the more symptomatic hand will be assigned to a shock wave treatment group, while the other hand will serve as a control. This means no treatment, but all measurements will be performed in the same way as in the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders
* aged above 18 years
* suffering from mild to moderate carpal tunnel syndrome with typical symptoms like pain, paresthesia, or fine motoric disorders:

  * very mild (grade 1): sensory nerve conduction velocity mildly reduced orslowercompared to the contralateral side.
  * mild (grade 2): distal motor latency <4,5ms and sensory nerve conduction velocity < 40 m/s
  * moderate (grade 3): distal motor latency between 4,5 and 6,5 ms and preserved sensory nerve amplitude.
* Patients with bilateral CTS also will be included, whereas the less symptomatic hand will be assessed as well, but receive no therapy.

Exclusion Criteria:

* Patients with severe CTS (distal motor latency above 6,5ms or absent sensory potentials);
* Prior therapy (even night splints) for CTS within the last six months
* The presence of common systemic diseases, that have known influence on the peripheral nerve system, like diabetes mellitus, polyneuropathy orabusive C2 consumption
* Postsurgical CTS
* Patients with serious injury of the wrist in medical history (e.g. radius fracture) or previous damage to median nerve and more proximal located compression syndrome of median nerve
* Patients with implanted electronic devices like defibrillators or pacemakers
* Pregnant women
* bifid median nerve;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | from enrollment until 32 weeks after first shockwave session
  The patient will be asked to categorize his pain and paresthesia on a numeric scale between 0 and 10.
Boston Carpal Tunnel Questionnaire | from enrollment until 32 weeks after first shockwave session
  Questionnaire to evaluate symptoms and functional restriction in daily activities in patients with CTS

SECONDARY OUTCOMES:
Nerve conduction study parameters | from enrollment until 32 weeks after first shockwave session
  Distal motor latency (DML):The electrode for assessingt he motoric fibers of the median nerve will be applied on the muscle belly of the thenar muscles. The orthodromic motoric stimulation will be performed 6,5 centimeters proxima l to the recording site at the height of the wrist with a single electric impulse. The time between stimulation and the initialincrease of the respondingcompoundm usclea ction potential (CMAP)i s namedt he DML.
Neurosonography of median nerve | from enrollment until 32 weeks after first shockwave session
  * Cross-sectional area (CSA): The cross-sectional area of the median nerve will be measured at a typical location at the height of the os pisiforme. The increase in CSA is a well-investigated finding in CTS patients with a cut-off value of about 10 mm2.
  * CSA differences: At the proximal third of the pronatorquadratus muscle (>10 centimeteß proximal) a second CSA measurement of the median nerve will be carried out. The difference between the proximal and the dista l values is also a specific and sensitive diagnostic criterion for CTS
Nerve conduction study parameters | from enrollment until 32 weeks after first shockwave session
  -Sensory nerve conduction velocity: A ring electrode (cathode) is placed on the index finger at the height of the proximal interphalangeal joint. The median nerve will be electrically stimulated antidromically at the same height on the wrist as in DML measurement (approximately 13-14 centimeters proximal to the recording site). For calculation of the nerve conduction velocity, the knowledge of the exact distance between the stimulation and the recording site of the nerve is necessary and therefore will be measure

IPD SHARING:
Plan to Share IPD: No